CLINICAL TRIAL: NCT01051466
Title: Neurobiological Correlates of Antidepressant Response After Duloxetine Hydrochloride Treatment in Subjects With Major Depressive Disorder
Brief Title: A Study of the Neurobiology of Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12875; F1J-US-HMGO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Major Depressive Disorder; Healthy Participants
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Healthy Participants (No Intervention)

INTERVENTIONS:
Drug: Duloxetine — 60 milligrams (mg) administered orally daily for 8 weeks then 60-120 mg if non remitter or 60 mg if remitter for 4 additional weeks
  Other Names: Cymbalta, LY248686
  Arms: Duloxetine

SUMMARY:
Previous research studies have shown that depression is associated with changes in structure and activity in different parts of the brain and that antidepressant medication can affect brain activity in different parts of the brain in individuals suffering from depression. The primary purpose of the study is to find out more about how the antidepressant medication duloxetine affects brain activity and structure in individuals with depression.

DETAILED DESCRIPTION:
This study will evaluate participants with depression before treatment is initiated and during treatment, and compare them to a control group of healthy participants. The aim will be to better understand both the neurobiology of depression and how the neurobiology changes in response to treatment of depression and the outcome of treatment. The study will include a variety of assessments of the neurobiology of depression including: scans of brain areas are involved in depression by looking at structures in the brain and how they work and blood tests and how these change in relation to several measures of depression severity.

ELIGIBILITY:
Inclusion Criteria:

Major Depressive Disorder (MDD) participants:

* Are right-handed
* Meet criteria for single episode or recurrent MDD, without psychotic features, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and confirmed by Structured Clinical Interview for DSM-IV-TR (SCID-IV), without co-morbid DSM-IV Axis I or II disorder at screening
* Be free of current antidepressant medication for a minimum of 6 weeks for fluoxetine treatment or of 4 weeks of other antidepressant treatment
* Have a 17-item Hamilton Depression Rating Scale (HAMD17) total score of ≥18 at screening, and baseline
* Women of child-bearing potential must have negative urine pregnancy tests prior to enrollment and agree to use a reliable method of birth control during the study

Healthy Participants

* Are right-handed
* Have a HAMD17 total score of <7 at screening and baseline and must not meet the criteria for MDD based on the SCID-IV

Exclusion Criteria:

MDD participants and healthy participants:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device
* Treatment within the last 30 days with a drug that has not received regulatory approval
* Have previously completed or withdrawn from this study or any other study investigating duloxetine
* Have a history of substance abuse or dependence within the past 6 months
* A positive urine drug screen for any substances of abuse or dependence
* Have any current DSM-IV-TR co-morbid Axis I or II disorder as determined by participant's history or investigator assessment
* Have any history of bipolar disorder, a primary psychotic disorder (schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder), known Alzheimer's disease or mental retardation, or obsessive-compulsive disorder as determined by participant's history or investigator assessment
* Pregnant women, women who are breast-feeding, or women of childbearing potential who are not using a medically accepted means of contraception when engaging in sexual intercourse or have been surgically sterilized
* Are judged by the investigator to have serious suicidal risk or risk of self-harm
* Have a history of recurrent self-mutilation or self-harm
* Have uncontrolled narrow-angle glaucoma
* Have been diagnosed with an acute liver injury (such as hepatitis) or severe cirrhosis (Child-Pugh Class C)
* Have end-stage renal disease, a prior renal transplant, current renal dialysis, or severe renal impairment
* Have abnormal thyroid-stimulating hormone (TSH) concentration
* Have had electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or vagus nerve stimulation (VNS) within the past year
* Initiating psychotherapy within 6 weeks prior to study entry or during study participation, stopping, or changing psychotherapy after study entry
* Have frequent and/or severe allergic reactions with multiple medications, or known allergic reactions to the study medication
* Known hypersensitivity to duloxetine or any of the inactive ingredients
* Lack of response of the current episode to two or more adequate courses of antidepressant therapy at a clinically appropriate dose for a minimum of 4 weeks or in the judgment of the investigator the participant meets criteria for treatment-resistant depression
* Known human immunodeficiency virus (HIV) and other medical disorders that are known to affect central nervous system (CNS) structures or function as assessed by the investigator (for example, CNS neoplasms, neurosyphilis)
* Have a medical illness, a clinically significant laboratory abnormality, or is taking a CNS active medication that, in the opinion of the investigator, might interfere with study participation (for example, is likely to require hospitalization) or that, in the opinion of the investigator, might interfere with the interpretation of the primary endpoint (for example, hypertension or diabetes)
* Are unwilling or unable to comply with the study procedures

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom, United Kingdom

REFERENCES:
- [Derived] Fu CH, Costafreda SG, Sankar A, Adams TM, Rasenick MM, Liu P, Donati R, Maglanoc LA, Horton P, Marangell LB. Multimodal functional and structural neuroimaging investigation of major depressive disorder following treatment with duloxetine. BMC Psychiatry. 2015 Apr 14;15:82. doi: 10.1186/s12888-015-0457-2. PMID 25880400

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: Duloxetine: Participants with major depressive disorder (MDD), who successfully completed screening, received 60 milligrams (mg) up to 120 mg orally, once daily (QD) for 12 weeks. The initial starting dose was 60 mg duloxetine QD for the first 8 weeks. Then, remitters [defined as participants with a 17-item Hamilton Depression Rating Scale (HAMD17) total score ≤7] continued on 60 mg duloxetine QD, while non-remitters (HAMD17 total score >7) could have their duloxetine dose flexed between 60 mg QD up to 120 mg QD, based on the clinical judgment of the Principal Investigator and tolerability of the participant to the dose. At study completion, participants could optionally complete a 2-week dose down-titration taper.
- Healthy Participants: Healthy participants: Participants who successfully completed screening, were matched by age, gender, and intelligence quotient (IQ) to participants with MDD. IQ was measured by the Wechsler Adult Intelligence Scale - Third United Kingdom Edition (WAIS-III UK). Healthy participants did not receive study drug.
Period: Overall Study
Arm/Group | Duloxetine | Healthy Participants
Started | 32 | 28
Completed | 24 | 23
Not Completed | 8 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Entry Criteria Not Met | 0 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Healthy Participants | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.21 (11.23) | 39.19 (9.41) | 39.74 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 19 | 14 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  White | 18 | 16 | 34
  Asian | 10 | 4 | 14
  Black | 4 | 8 | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12-Week Endpoint in the Functional Magnetic Resonance Imaging (fMRI) Mean Blood Oxygenation-Level-Dependent (BOLD) Response in the Amygdalae
Description: Functional MRI or fMRI is a functional neuroimaging procedure that uses MRI technology to measure brain activity by detecting associated changes in blood flow. When an area of the brain is in use, blood flow to that region increases. The activation in response to the processing of sad faces was measured by the percentage of signal change in BOLD response from before to after sad faces processing. The percentage of signal change was calculated by taking the difference between BOLD response after sad faces processing and BOLD response before sad faces processing and dividing by BOLD response before sad face processing, then multiplying by 100. BOLD signals were measured using arbitrary magnetic resonance units. Amygdala BOLD activation was calculated as an average between the left amygdala activation and right amygdala activation. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline activation (BOLD response) observation.
Measure: Least Squares Mean (Standard Error); unit: percentage of signal change
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 28 | 28
percentage of signal change | -0.01 (0.13) | -0.16 (0.13)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.457, Mixed Models Analysis — The significance level was 0.05 for a 2-sided test

2. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Activation [Blood Oxygenation-Level-Dependent (BOLD) Response to Implicit Processing of Sad Faces] for Each of the 3 Brain Regions
Description: Functional magnetic resonance imaging (fMRI) is a functional neuroimaging procedure that uses MRI technology to measure brain activity by detecting associated changes in blood flow. When an area of the brain is in use, blood flow to that region increases. The activation in response to the processing of sad faces in each brain region (anterior cingulate, left amygdala and right amygdala) was measured by the percentage of signal change in BOLD response. The percentage of signal change was calculated by taking the difference between BOLD response after sad faces processing and BOLD response before sad faces processing and dividing by BOLD response before sad face processing, then multiplying by 100. BOLD signals were measured using arbitrary magnetic resonance units. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline activation (BOLD response) observation, excluding 3 healthy participants who did not meet entry criteria.
Measure: Least Squares Mean (Standard Error); unit: percentage of signal change
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 28 | 25
percentage of signal change
  Anterior Cingulate | 0.13 (0.09) | 0.20 (0.09)
  Left Amygdala | -0.04 (0.16) | -0.26 (0.16)
  Right Amygdala | 0.03 (0.12) | -0.09 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.627, Mixed Models Analysis — The p-value is for change from baseline activation (BOLD response) in the anterior cingulate
Statistical Analysis 2: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.338, Mixed Models Analysis — The p-value is for change from baseline activation (BOLD response) in the left amygdala
Statistical Analysis 3: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.518, Mixed Models Analysis — The p-value is for change from baseline activation (BOLD response) in the right amygdala

3. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Volume of Subgenual Anterior Cingulate, Amygdalae, and Hippocampus
Description: The volume of specific brain regions is obtained using a structural magnetic resonance imaging (sMRI) procedure in which high-resolution spoiled gradient recall images are acquired in coronal brain slices. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline observation for the volume of specific brain regions, excluding 3 healthy participants who did not meet entry criteria.
Measure: Least Squares Mean (Standard Error); unit: cubic millimeters (mm^3)
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 28 | 24
cubic millimeters (mm^3)
  Subgenual Anterior Cingulate | -188.27 (112.37) | 175.22 (116.14)
  Left Amygdalae | -23.68 (15.25) | 4.20 (15.59)
  Right Amygdalae | -33.38 (17.83) | 23.86 (18.40)
  Left Hippocampus | -13.56 (23.53) | 18.52 (24.37)
  Right Hippocampus | -14.70 (19.19) | 21.80 (19.66)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — The p-value is for change from baseline volume in the subgenual anterior cingulate
Statistical Analysis 2: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.208, Mixed Models Analysis — The p-value is for change from baseline volume in the left amygdalae
Statistical Analysis 3: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.031, Mixed Models Analysis — The p-value is for change from baseline volume in the right amygdalae
Statistical Analysis 4: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.350, Mixed Models Analysis — The p-value is for change from baseline volume in the left hippocampus
Statistical Analysis 5: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.191, Mixed Models Analysis — The p-value is for change from baseline volume in the right hippocampus

4. Secondary Outcome: Translocation of Gs Alpha (Gsα) From Lipid Rafts in the Cell Membranes of Red Blood Cells (RBCs), White Blood Cells (WBCs) and Platelets Compared With Baseline
Description: Gsα is a membrane-associated protein that couples receptors for neurotransmitters like serotonin to allow them to send messages between nerve cells - a process that may be altered during depression and antidepressant treatment. Gsα localization in the cholesterol-rich (lipid rafts) and cholesterol-poor regions of cell membranes of RBCs and platelets was measured with quantitative Western blots and reported as the ratio of Gsα (absorbance units) in Triton X-100 (TX-100) over Triton X-114 (TX-114), 2 detergents that discriminate between lipid raft and non-raft membrane domains. Translocation of Gsα was measured as the change from baseline in Gsα localization. Translocation of Gsα from lipid rafts in the cell membranes of WBCs was not analyzed due to technical laboratory issues. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Weeks 1, 8, and 12
Population: Enrolled participants who had a baseline and at least 1 post-baseline Gsα localization observation, excluding 3 healthy participants who did not meet entry criteria. No participants were analyzed for the translocation of Gsα from lipid rafts in the cell membranes of WBCs.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 23 | 22
Ratio
  RBCs, Week 1 (n=23, 22) | 0.51 (0.21) | 0.09 (0.22)
  RBCs, Week 8 (n=23, 22) | -0.01 (0.14) | -0.15 (0.14)
  RBCs, Week 12 (n=23, 22) | 0.36 (0.26) | 0.10 (0.26)
  Platelets, Week 1 (n=23, 20) | -0.63 (0.46) | -0.69 (0.49)
  Platelets, Week 8 (n=23, 20) | -1.16 (0.42) | -0.92 (0.44)
  Platelets, Week 12 (n=23, 20) | -0.52 (5.40) | 7.93 (5.40)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.174, Mixed Models Analysis — The p-value is for Gsα translocation in RBCs at Week 1
Statistical Analysis 2: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.488, Mixed Models Analysis — The p-value is for Gsα translocation in RBCs at Week 8
Statistical Analysis 3: Comparison: Healthy Participants; Test type: Superiority or Other; p = 0.480, Mixed Models Analysis — The p-value is for Gsα translocation in RBCs at Week 12
Statistical Analysis 4: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.925, Mixed Models Analysis — The p-value is for Gsα translocation in platelets at Week 1
Statistical Analysis 5: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.697, Mixed Models Analysis — The p-value is for Gsα translocation in platelets at Week 8
Statistical Analysis 6: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.276, Mixed Models Analysis — The p-value is for Gsα translocation in platelets at Week 12

5. Secondary Outcome: Gs Alpha (Gsα)-Activated Adenylyl Cyclase
Description: Gsα is a membrane-associated protein that couples receptors for neurotransmitters like serotonin to allow them to send messages between nerve cells - a process that may be altered during depression and antidepressant treatment. Adenylyl cyclase is activated by Gsα, and when Gsα is translocated from lipid rafts it more effectively activates adenylyl cyclase. Gsα-activated adenylyl cyclase was not analyzed due to technical laboratory issues.
Time Frame: Baseline and Weeks 1, 8, and 12
Population: No participants were analyzed.
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Brain-Derived Neurotrophic Factor (BDNF) and the Precursor of BDNF (proBDNF)
Description: There is evidence that stress may decrease BDNF expression, while antidepressant treatment reverses or blocks these effects. BDNF is a protein that occurs naturally and supports the survival and growth of some nerve cells in the brain. proBDNF is a precursor of BDNF. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline BDNF or proBDNF observation, excluding 3 healthy participants who did not meet entry criteria.
Measure: Least Squares Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 23 | 21
nanograms per milliliter (ng/mL)
  BDNF (n=23, 21) | 6.61 (23.38) | 10.57 (22.80)
  proBDNF (n=13, 17) | -5.67 (12.77) | -9.37 (9.36)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.904, Mixed Models Analysis — The p-value is for change from baseline BDNF
Statistical Analysis 2: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.819, Mixed Models Analysis — The p-value is for change from baseline proBDNF

7. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Brain-Derived Neurotrophic Factor (BDNF) and the Precursor of BDNF (proBDNF) Receptors
Description: There is evidence that stress may decrease BDNF expression, while antidepressant treatment reverses or blocks these effects. BDNF is a protein that occurs naturally and supports the survival and growth of some nerve cells in the brain. proBDNF is a precursor of BDNF. Tropomyosin receptor kinase B (trkB) is a receptor for BDNF, and pan-neurotrophin receptor p75 (p75NTR) is a receptor for proBDNF. p75NTR was not analyzed due to technical laboratory issues. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline trkB observation, excluding 3 healthy participants who did not meet entry criteria. No participant was analyzed for the change from baseline in p75NTR receptors.
Measure: Least Squares Mean (Standard Error); unit: picograms per milligram (pg/mg)
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 24 | 21
picograms per milligram (pg/mg) | 52.1 (41.08) | -8.9 (36.25)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.273, Mixed Models Analysis — The p-value is for change from baseline trkB

8. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Proinflammatory Cytokines [Tumor Necrosis Factor Alpha (TNFα), Interleukin 1 (IL-1), and Interleukin 6 (IL-6)]
Description: Cytokines are naturally produced and regulate responses to inflammation. Proinflammatory cytokines like TNFα, IL-1, and IL-6 increase inflammation in the body. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) adjusted for group, visit, group-by-visit, and baseline value.
Time Frame: Baseline, Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline cytokine observation (TNFα, IL-1, or IL-6), excluding 3 healthy participants who did not meet entry criteria.
Measure: Least Squares Mean (Standard Error); unit: picograms per milliliter (pg/mL)
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 28 | 22
picograms per milliliter (pg/mL)
  Cytokine TNFα | -0.04 (0.78) | 0.25 (0.81)
  Cytokine IL-1 | -0.08 (2.53) | 4.01 (2.64)
  Cytokine IL-6 | -0.61 (0.69) | -0.52 (0.71)
Statistical Analysis 1: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.797, Mixed Models Analysis — The p-value is for change from baseline cytokine TNFα
Statistical Analysis 2: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.269, Mixed Models Analysis — The p-value is for change from baseline cytokine IL-1
Statistical Analysis 3: Comparison: Duloxetine vs Healthy Participants; Test type: Superiority or Other; p = 0.925, Mixed Models Analysis — The p-value is for change from baseline cytokine IL-6

9. Secondary Outcome: 17-Item Hamilton Depression Rating Scale (HAMD17)
Description: The HAMD17 is a standardized instrument consisting of 17 items used to measure the severity of major depressive disorder (MDD) and improvements in depression symptoms. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicated greater symptom severity. The total score was the sum of the scores from HAMD17 Items 1 through 17 and could have ranged from 0 (not at all depressed) to 52 (severely depressed).
Time Frame: Baseline and up to Week 12
Population: Enrolled participants who had a baseline and at least 1 post-baseline HAMD17 observation. Last observation carried forward (LOCF) was utilized when calculating the Week 12 endpoint outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 29 | 14
units on a scale
  Baseline | 22.4 (2.66) | 0.5 (1.34)
  Week 12 | 8.5 (6.60) | 0.5 (1.40)

10. Secondary Outcome: Percentage of Participants With 17-Item Hamilton Depression Rating Scale (HAMD17) Response
Description: HAMD17 response is defined as a >50% reduction in HAMD17 total score from baseline. The HAMD17 is a standardized instrument consisting of 17 items used to measure the severity of major depressive disorder (MDD) and improvements in depression symptoms. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicated greater symptom severity. The total score was the sum of the scores from HAMD17 Items 1 through 17 and could have ranged from 0 (not at all depressed) to 52 (severely depressed). The percentage of participants with a HAMD17 response was calculated as the number of participants with a >50% reduction in HAMD17 total score from baseline divided by the number of participants who had a HAMD17 observation at Week 12 then multiplied by 100.
Time Frame: Baseline, up to Week 12
Population: Enrolled MDD participants who had a baseline and at least 1 post-baseline HAMD17 observation. Last observation carried forward (LOCF) was utilized when calculating the Week 12 endpoint outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 29
percentage of participants | 72.4

11. Secondary Outcome: Percentage of Participants With 17-Item Hamilton Depression Rating Scale (HAMD17) Remission
Description: HAMD17 remission is defined as a HAMD17 total score of ≤7 at Week 12 (endpoint). The HAMD17 is a standardized instrument consisting of 17 items used to measure the severity of major depressive disorder (MDD) and improvements in depression symptoms. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicated greater symptom severity. The total score was the sum of the scores from HAMD17 Items 1 through 17 and could have ranged from 0 (not at all depressed) to 52 (severely depressed). The percentage of participants with remission was calculated as the number of participants with a HAMD17 total score of ≤7 divided by the number of participants who had a HAMD17 observation at Week 12 then multiplied by 100.
Time Frame: Baseline, up to Week 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 29
percentage of participants | 62.1

12. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The SDS is a participant-rated questionnaire used to assess the effect of the participant's symptoms on work/school (Item 1), social life/leisure activities (Item 2), and family/home management (Item 3). Each item was rated on a visual analog scale (VAS) from 0 (not at all) to 10 (very severely). The SDS Global Functional Impairment Score (SDS Global Score) was the sum of the 3 items and could have ranged from 0 (unimpaired) to 30 (highly impaired). Higher values indicated higher functional impairment in the participant's work/social/family life.
Time Frame: Baseline and up to Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline SDS observation. Last observation carried forward (LOCF) was utilized when calculating the Week 12 endpoint outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Healthy Participants: Healthy participants: Participants who successfully completed screening were matched by age, gender, and intelligence quotient (IQ) to participants with MDD. IQ was measured by the Wechsler Adult Intelligence Scale - Third United Kingdom Edition (WAIS-III UK). Healthy participants did not receive study drug.
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 27 | 25
units on a scale
  Baseline | 19.3 (5.41) | 0.2 (0.80)
  Week 12 | 9.4 (7.72) | 0.0 (0.00)

13. Secondary Outcome: Clinical Global Impressions of Severity Scale (CGI-S)
Description: The CGI-S measures severity of illness at the time of assessment. Scores can range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline and up to Week 12
Population: Enrolled participants who had baseline and at least 1 post-baseline CGI-S observation. Last observation carried forward (LOCF) was utilized when calculating the Week 12 endpoint outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 29 | 25
units on a scale
  Baseline | 4.4 (0.56) | 1.0 (0.00)
  Week 12 | 2.2 (1.08) | 1.0 (0.00)

14. Secondary Outcome: Patient's Global Impressions of Improvement (PGI-I) Scale
Description: The PGI-I scale measures the participant's perception of improvement at the time of assessment compared with the start of treatment. Scores can range from 1 (very much better) to 7 (very much worse).
Time Frame: Baseline, up to Week 12
Population: Enrolled MDD participants who had at least 1 post-baseline PGI-I observation. Last observation carried forward (LOCF) was utilized when calculating the Week 12 endpoint outcome. PGI-I observations were not completed for healthy participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 29
units on a scale | 2.6 (1.24)

15. Secondary Outcome: Hamilton Anxiety Rating Scale (HAMA)
Description: The 14-item HAMA is used to assess the severity of anxiety. The investigator talked to the participant about their symptoms over the previous week. Each item was scored using a 5-point scale (0 = not present to 4 = very severe). Total HAMA scores could have ranged from 0 (normal) to 56 (severe).
Time Frame: Baseline and up to Week 12
Population: Enrolled participants who had a baseline and at least 1 post-baseline HAMA observation. Last observation carried forward (LOCF) was utilized when calculating the Week 12 endpoint outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Healthy Participants: Healthy participants: Participants who successfully completed screening were matched by age, gender, and intelligence quotient (IQ) to participants with MDD. IQ was measured by the Wechsler Adult Intelligence Scale - Third United Kingdom (UK) Edition (WAIS-III^UK). Healthy participants did not receive study drug.
Arm/Group | Duloxetine | Healthy Participants
Number analyzed (Participants) | 29 | 25
units on a scale
  Baseline | 21.1 (5.78) | 0.4 (0.87)
  Week 12 | 9.6 (7.25) | 0.4 (0.96)

16. Secondary Outcome: Incidence of Suicidal Behavior and Suicidal Ideation as Measured by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captures the occurrence, severity, and frequency of treatment-emergent suicide-related thoughts and behaviors. Suicidal ideation is defined as a "yes" answer to any 1 of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior is defined as a "yes" answer to any 1 of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Treatment-emergent outcomes were the worsening or new occurrence of suicidal behaviors or ideation during treatment compared with baseline.
Time Frame: Baseline through Week 12
Population: Participants with MDD who had a baseline and at least 1 post-baseline C-SSRS assessment. Healthy participants did not have a C-SSRS assessment post baseline.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 29
participants
  Treatment-emergent suicidal ideation | 5
  Treatment-emergent suicidal behavior | 0

ADVERSE EVENTS:
Groups:
- Duloxetine: Duloxetine: Participants with major depressive disorder (MDD) received 60 milligrams (mg) up to 120 mg orally, once daily (QD) for 12 weeks. The initial starting dose was 60 mg duloxetine QD for the first 8 weeks. Then, remitters [defined as participants with a 17-item Hamilton Depression Rating Scale (HAMD17) total score ≤7] continued on 60 mg duloxetine QD, while non-remitters (HAMD17 total score >7) could have their duloxetine dose flexed between 60 mg QD up to 120 mg QD, based on the clinical judgment of the Principal Investigator and tolerability of the participant to the dose.
- Healthy Participants: Healthy participants: Participants were matched by age, gender, and intelligence quotient (IQ) to participants with MDD. IQ was measured by the Wechsler Adult Intelligence Scale - Third United Kingdom Edition (WAIS-III UK). Healthy participants did not receive study drug.
Arm/Group | Duloxetine | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/28
Other Adverse Events (participants affected / at risk) | 32/32 | 11/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=32) | Healthy Participants (N=28)
Retinal pigment epitheliopathy (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine (N=32) | Healthy Participants (N=28)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (23) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sluggishness (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (7) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Gastric ph decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 0 (0)
Food craving (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 9 (11) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 11 (18) | 4 (8)
Hypersomnia (Nervous system disorders) | 2 (2) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 4 (5) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
White matter lesion (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Anorgasmia (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (9) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Ejaculation delayed (Reproductive system and breast disorders) | 1/19 (1) | 0/14 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 1/19 (1) | 0/14 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/19 (1) | 0/14 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Yawning (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Three healthy participants were identified as not meeting inclusion/exclusion criteria after enrollment. They were discontinued and excluded from secondary outcome analyses, but included in participant flow, primary outcome analyses, and safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days